CLINICAL TRIAL: NCT00855322
Title: Randomized Controlled Trial Examining The Effect Of Exercise In People With Rheumatoid Arthritis Taking Anti-TNFalpha Medication
Brief Title: Study Examining the Effect of Exercise in People With Rheumatoid Arthritis Taking Anti-TNFalpha Medication
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College Dublin (Other)
Responsible Party: Dr Tara Cusack, University College Dublin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RAEx-0809
Record Dates: First submitted 2009-03-02; First posted 2009-03-04 (Estimated); Last update posted 2009-03-04 (Estimated); Status verified 2009-02

CONDITIONS: Arthritis, Rheumatoid
Keywords: Arthritis, Rheumatoid; Exercise; Biological Therapy
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Gym group exercise intervention
  Interventions: Other: Gym exercise group intervention
- 2 (Experimental): Hydrotherapy group exercise intervention
  Interventions: Other: Hydrotherapy group exercise intervention
- 3 (No Intervention): Control group
  Interventions: Other: Control group

INTERVENTIONS:
Other: Gym exercise group intervention — Gym based circuit class
  Other Names: Gym Group
  Arms: 1
Other: Hydrotherapy group exercise intervention — Hydrotherapy group exercise class
  Other Names: Aquatic Physiotherapy
  Arms: 2
Other: Control group — No intervention
  Arms: 3

SUMMARY:
The purpose of this study is to determine whether exercise is beneficial for people with rheumatoid arthritis(RA) taking antiTNFalpha medication

DETAILED DESCRIPTION:
Substantial progress has been made in the medical management of RA over the past decade but at present no drug therapy leads to long-term remission for all patients with RA. People may still continue to experience physical, psychological and functional consequences which could benefit from rehabilitation.little research exists on the effects of exercise for people with RA taking anti-TNFalpha therapy medication.

It is proposed to conduct a randomized controlled trial to examine the effects of group exercise therapy in a gym setting or in a hydrotherapy pool compared to a control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with RA receiving anti-TNFalpha therapy medication for more than three months
* Consenting male and female patients aged 18 - 70 years
* Patients will have a documented diagnosis of RA as classified by the American College of Rheumatology (ACR) criteria
* ACR functional class I, II, III

Exclusion Criteria:

* Patients who have attended physiotherapy in the past three months
* Patients to whom exercise therapy or hydrotherapy are contraindicated
* Patients who have undergone joint surgery in the past six months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-07 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
Stanford Health Assessment Questionnaire | Baseline, 8 weeks and 24 weeks

SECONDARY OUTCOMES:
50 foot Walk Test | Baseline, 8 weeks and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Oliver FitzGerald, MB, BcH, BAO, Principal Investigator — University College Dublin; Tara Cusack, PhD, MMedSc,, Study Director — University College Dublin
Locations (1):
- Our Lady's Hospice, Dublin, Dublin, Ireland

REFERENCES:
- [Derived] Reid A, Brady A, Blake C, Mongey AB, Veale DJ, FitzGerald O, Cusack T. Randomised controlled trial examining the effect of exercise in people with rheumatoid arthritis taking anti-TNFalpha therapy medication. BMC Musculoskelet Disord. 2011 Jan 13;12:11. doi: 10.1186/1471-2474-12-11. PMID 21232112